CLINICAL TRIAL: NCT04655131
Title: Effect of Protein Intake on Post Prandial Hyperglycemia in Children and Adolescents With Type1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Dalia Dalle, Primary investigator, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-18-18
Record Dates: First submitted 2020-11-22; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 1; Hyperglycemia, Postprandial
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Protein consumption : 0 gm (Active Comparator): Participant's glucose levels are monitored from hour 0 to hour 5 after consumption of 0 gm of whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate
- Protein consumption : 12.5 gm (Experimental): Participant's glucose levels are monitored from hour 0 to hour 5 after consumption of 12.5 gm of whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate
- Protein consumption : 25 gm (Experimental): Participant's glucose levels are monitored from hour 0 to hour 5 after consumption of 25 gm of whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate
- Protein consumption :37.5 gm (Experimental): Participant's glucose levels are monitored from hour 0 to hour 5 after consumption of 37.5 gm of whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate
- Protein consumption : 50 gm (Experimental): Participant's glucose levels are monitored from hour 0 to hour 5 after consumption of 50 gm of whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate
- Protein consumption : 62.5 gm (Experimental): Participant's glucose levels are monitored from hour 0 to hour 5 after consumption of 62.5 gm of whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate

INTERVENTIONS:
Dietary Supplement: Whey protein isolate — Commercially available, FDA approved whey protein isolate for dietary supplementation

SUMMARY:
In type 1 Diabetes Mellitus, patients receive insulin doses if they consume specific amounts of carbohydrates. Currently, insulin is not being administered for consumption of protein although studies in adults show that consuming about 75 grams of protein causes elevation in post prandial glucose levels and might need insulin coverage. We are proposing that this amount is different for kids and it might vary based on weight, age, pubertal stage, HbA1C or other factors.

This has not been studied in children before, and it will provide information about the amount of protein in the diet that can cause elevation in post prandial glucose.

DETAILED DESCRIPTION:
In target glycemic control in children with type 1 diabetes (T1D) continues to be a challenge despite advances in methods of insulin delivery and medical knowledge in this area. One of the major aspects is controlling postprandial glycemia (PPG). The relationship between dietary intake of carbohydrates and PPG is well established, and the use of insulin coverage for carbohydrate intake is standard of care. Insulin dose for carbohydrate coverage increases with body weight and progression through puberty. Multiple researchers have attempted to study the effect of dietary intake of protein and fat on PPG as well, but this relationship is not well established in the pediatric age group and there are not clear guidelines for patients on when and how to give insulin for protein intake.

Meals with high protein content have been shown to cause higher glucose excursions in patients with T1D, and lower glycemic response in healthy individuals which suggests that physiologic response to protein intake involves higher insulin secretion. This has also been demonstrated by Sun et al, where they showed an increase in insulinemic index in healthy individuals when consuming chicken with rice compared to rice alone.

The effect of dietary protein in individuals with T1D has been studied in mixed meals several times. Smart et al demonstrated that the greatest glucose excursions after high protein low fat meal occurred most significantly form min 150 to 300 after the meal, when insulin is given to cover carbohydrates only. In 2013, Borie-Swinburne et al measured interstitial glucose levels by CGM in 28 c-peptide negative T1D patients, on two consecutive nights, with and without addition of 21.5 grams of protein to dinner (40 g vs 61.5 g). They concluded that no additional insulin is needed to cover for the added protein. Neu et al studied 15 adolescents with T1D on two consecutive nights. They used CGM monitoring for 12 hours, and they compared the area under the curve (AUC) between regular meals and fat/ protein rich meal. They found a significant difference and they recommended additional insulin for fat /protein rich meals.

Investigating the effect of protein-only intake is also an area of research focus. Paterson et al studied 27 patients with TID , aged 7-40 yrs, where they were given 6 test meals of varying amounts (0g, 12.5g, 25g, 50g, 75g and 100g) of pure protein without giving insulin. Postprandial glycemia was found to be significantly higher only for 75 and 100 grams of protein compared to the lower quantities. Glucose levels were slower to rise when compared to consumption of 20 grams of carbohydrates. Paterson et al also conducted another study with slightly different design: 27 participants with T1D [aged 10-40 years, HbA1c ≤ 64 mmol/mol (8%), BMI ≤ 91st percentile] received a 30-g carbohydrate (negligible fat) test drink with a variable amount of protein daily over 5 days in randomized order. Protein (whey isolate 0 g/kg carbohydrate, 0 g/kg lipid) was added in amounts of 0 (control), 12.5, 25, 50 and 75 g. A standardized dose of insulin was given for the carbohydrate. PPG was assessed by 5 hours of continuous glucose monitoring. Increasing protein quantity in a low-fat meal containing consistent amounts of carbohydrate decreases glucose excursions in the early (0-60-min) postprandial period and then increases in the later postprandial period in a dose-dependent manner. In summary, Paterson et al concluded that there was a threshold for dietary protein intake (75 grams), and only protein intake above this threshold regardless of body weight would result in post prandial hyperglycemia. However, these studies included a wide range of ages and did not adjust for body weight in their analysis.

B. Innovation The purpose of this study is to explore the role of weight in the relationship between protein intake and post prandial glucose (PPG) levels. The study design (36 children each receiving 6 increasing nominal doses of protein) allows for the relationship to be studied both across patients of varying weights within each nominal dose, and across patients (whose weights remain the same) across the increasing doses.

Our aims:

Aim 1: To describe the relationship of weight (in kg), and mg of protein per kg body weight, to PPG, graphically and statistically, at each nominal dose. The heaviest children will receive the lowest mg/kg amount of protein at each nominal dose, so these relationships with PPG will be inverse. Additionally, children with different weights and receiving different nominal doses, may be receiving the same mg/kg protein. Observing all nominal doses together will allow us to determine whether the relationship, if any, is linear, demonstrates a threshold, or exhibits a doseresponse curve, as examples.

Aim 2: To describe graphically and statistically the relationship of dose of protein to PPG by patient across increasing doses. Since the weight remains constant (or approximately constant) within a patient, adjustment by weight would yield the same results. The expectation is that these results will confirm those from Aim 1.

Aim 3: To construct a multivariate mixed model where any observed relationships can be controlled for other demographic and clinical characteristics possibly associated with blood glucose levels. The type of model will depend on the results of Aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

. Duration of type 1 diabetes for > 1year.

* On insulin pump or multiple daily injection regimen
* Uses a personal Dexcom CGM
* Age: 5- 17 years
* HbA1C range: < 9%

Exclusion Criteria:

* Hyperlipidemia
* Diabetic gastroparesis
* Dietary restrictions
* Celiac disease and other malabsorption syndromes
* Uncontrolled hypothyroidism
* Chronic use of steroids or antipsychotics
* Metabolic disorders of gluconeogenesis
* Use of oral hypoglycemic agents
* Participating in another clinical trial

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Number of positive events for each protein amount. | from hour 0 to hour 5 after intervention
  Events of postprandial hyperglycemia were defined as rise in glucose >50 mg/dL compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Dalle, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04655131/Prot_SAP_000.pdf